CLINICAL TRIAL: NCT02966795
Title: A Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Glecaprevir (GLE)/Pibrentasvir (PIB) in Adults With Chronic Hepatitis C Virus (HCV) Genotype 5 or 6 Infection
Brief Title: A Study of of Glecaprevir/Pibrentasvir in Adults With Chronic Hepatitis C Virus (HCV) Genotype 5 or 6 Infection
Acronym: ENDURANCE-5 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-126; 2016-003192-22 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: glecaprevir; pibrentasvir; compensated cirrhosis; non-cirrhotic; interferon (IFN); pegylated interferon (pegIFN); ribavirin (RBV); sofosbuvir (SOF); Sustained Virologic Response 12 weeks post dosing (SVR12); Chronic; Genotype 5 or 6 Infection
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glecaprevir/Pibrentasvir for 8 Weeks (Experimental): Non-cirrhotic participants with hepatitis C virus genotype 5 or 6 received oral glecaprevir/pibrentasir (300 mg/120 mg) once daily with food for 8 weeks, according to label.
  Interventions: Drug: Glecaprevir/Pibrentasvir
- Glecaprevir/Pibrentasvir for 12 Weeks (Experimental): Participants with hepatitis C virus genotype 5 or 6 and compensated cirrhosis received oral glecaprevir/pibrentasir (300 mg/120 mg) once daily with food for 12 weeks, according to label.
  Interventions: Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir — Fixed-dose combination tablets taken orally once a day.
  Other Names: ABT-493/ABT-530; MAVYRET™

SUMMARY:
A Phase 3b, open-label, multicenter study to evaluate the efficacy and safety of glecaprevir/pibrentasvir for an 8- or 12-week treatment duration in participants with chronic hepatitis C virus (HCV) genotype (GT) 5 or 6 infection, with or without compensated cirrhosis respectively.

ELIGIBILITY:
Inclusion Criteria:

* Screening laboratory result indicating hepatitis C virus (HCV) GT5 or 6 infection.
* Participant has a positive anti-HCV antibody (Ab) and plasma HCV ribonucleic acid (RNA) greater than or equal to 1000 IU/mL at Screening Visit.
* Participant must be HCV treatment-naïve (i.e., has never received a single dose of any approved or investigational anti-HCV medication) or treatment-experienced (i.e., has failed prior interferon [IFN] or pegylated interferon [pegIFN] with or without ribavirin [RBV], or sofosbuvir [SOF] plus RBV with or without pegIFN therapy). Prior HCV treatment with any other approved or investigational medications is not allowed. Previous HCV treatment must have been completed greater than or equal to 2 months prior to screening.
* Participant must be documented as having no cirrhosis or compensated cirrhosis.

Exclusion Criteria:

* Female participant who is pregnant, breastfeeding, or is considering becoming pregnant during the study or for approximately 30 days after the last dose of study drug.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
* HCV genotype performed during screening indicating co-infection with more than one HCV genotype.
* History of severe, life-threatening or other significant sensitivity to any excipients of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (25):
- United States (6):
  - Research & Education, Inc. /ID# 157042, San Diego, California
  - Kaiser Permanente /ID# 157044, San Diego, California
  - Zuckerberg San Francisco Gener /ID# 157040, San Francisco, California
  - Cedars-Sinai Medical Center - West Hollywood /ID# 157045, West Hollywood, California
  - Einstein Medical Center /ID# 157436, Philadelphia, Pennsylvania
  - University of Washington /ID# 157041, Seattle, Washington
- Australia (3):
  - Nepean Hospital Kingswood /ID# 157027, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 157025, Herston, Queensland
  - Royal Melbourne Hospital /ID# 157024, Parkville, Victoria
- Belgium (2):
  - AZ Groeninge /ID# 157029, Kortrijk
  - UZ Leuven /ID# 157030, Leuven
- Canada (2):
  - University of Calgary /ID# 157031, Calgary, Alberta
  - Toronto General Hospital /ID# 157032, Toronto, Ontario
- France (4):
  - Hopital Haut-Lévêque /ID# 157035, Pessac, Gironde
  - CHU Estaing /ID# 157034, Clermont-Ferrand
  - Hopital Saint Antoine /ID# 157036, Paris
  - Hopital Beaujon /ID# 157028, Clichy, Île-de-France Region
- Auckland Clinical Studies Ltd /ID# 157033, Auckland, New Zealand
- Singapore (2):
  - National University Hospital /ID# 156855, Singapore
  - Singapore General Hospital /ID# 157037, Singapore
- South Africa (2):
  - Wits Clinical Research Site /ID# 157038, Johannesburg, Gauteng
  - University of Cape Town /ID# 157039, Cape Town, Western Cape
- Vietnam (3):
  - National Hospital of Tropical Diseases /ID# 162282, Hanoi
  - Hoa Hao Medic Co. Ltd. /ID# 162283, Ho Chi Minh City
  - Tropical Diseases Hospital /ID# 162281, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Asselah T, Lee SS, Yao BB, Nguyen T, Wong F, Mahomed A, Lim SG, Abergel A, Sasadeusz J, Gane E, Zadeikis N, Schnell G, Zhang Z, Porcalla A, Mensa FJ, Nguyen K. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic hepatitis C virus genotype 5 or 6 infection (ENDURANCE-5,6): an open-label, multicentre, phase 3b trial. Lancet Gastroenterol Hepatol. 2019 Jan;4(1):45-51. doi: 10.1016/S2468-1253(18)30341-8. Epub 2018 Nov 2. PMID 30393106
- [Derived] Brown RS Jr, Collins MA, Strasser SI, Emmett A, Topp AS, Burroughs M, Ferreira R, Feld JJ. Efficacy and Safety of 8- or 12 Weeks of Glecaprevir/Pibrentasvir in Patients with Evidence of Portal Hypertension. Infect Dis Ther. 2022 Apr;11(2):913-924. doi: 10.1007/s40121-022-00599-8. Epub 2022 Feb 17. PMID 35174470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 24 hospitals or clinics in Europe (Belgium, France), Oceania (Australia, New Zealand), North America (Canada, USA), South Africa, and southeast Asia (Singapore, Vietnam). Participants were screened between January 17, 2017, and December 26, 2017.
Pre-assignment Details: Enrolled participants with genotype 5 or 6 hepatitis C (HCV) were assigned to treatment with glecaprevir/pibrentasir for either 8 weeks or 12 weeks based on cirrhotic status.
Groups:
- Genotype 5-infected: Participants with HCV genotype 5 infection received oral glecaprevir/pibrentasir (300 mg/120 mg) once daily with food for either 8 weeks (those without cirrhosis) or 12 weeks (those with compensated cirrhosis), according to label.
- Genotype 6-infected: Participants with HCV genotype 6 infection received oral glecaprevir/pibrentasir (300 mg/120 mg) once daily with food for either 8 weeks (those without cirrhosis) or 12 weeks (those with compensated cirrhosis), according to label.
Period: Overall Study
Arm/Group | Genotype 5-infected | Genotype 6-infected
Started | 23 | 61
Completed | 23 | 60
Not Completed | 0 | 1
Not completed — Patient Left the Country | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Genotype 5-infected; Genotype 6-infected: Participants received oral glecaprevir/pibrentasir (300 mg/120 mg) once daily with food for either 8 weeks (those without cirrhosis) or 12 weeks (those with compensated cirrhosis), according to label.
- Total: Total of all reporting groups
Arm/Group | Genotype 5-infected | Genotype 6-infected | Total
Number analyzed (Participants) | 23 | 61 | 84
Age, Continuous [Median (Full Range); unit: years] | 68.0 [24 to 76] | 54.0 [30 to 79] | 59.0 [24 to 79]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 8 | 45 | 53
  ≥ 65 years | 15 | 16 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 32 | 45
  Male | 10 | 29 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 61 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 4 | 25
  Black or African American | 1 | 0 | 1
  Asian | 1 | 56 | 57
  Multi-race | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 3 | 4
  Canada | 0 | 13 | 13
  Vietnam | 0 | 12 | 12
  Singapore | 0 | 4 | 4
  Belgium | 8 | 0 | 8
  United States | 0 | 15 | 15
  South Africa | 3 | 1 | 4
  Australia | 0 | 8 | 8
  France | 11 | 5 | 16
Cirrhosis Status [Count of Participants; unit: Participants]
  Cirrhotic | 3 | 6 | 9
  Non-cirrhotic | 20 | 55 | 75
Prior HCV Treatment History [Count of Participants; unit: Participants]
  Naive | 19 | 57 | 76
  Experienced | 4 | 4 | 8
HCV Ribonucleic Acid (RNA) Concentration [Mean (Standard Deviation); unit: log10 IU/mL] | 6.52 (0.53) | 6.64 (0.74) | 6.61 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post Treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ; less than 15 IU/mL) 12 weeks after the last actual dose of study drug.
Time Frame: 12 weeks after last dose of study drug (week 20 or 24 depending on the treatment regimen)
Population: All enrolled participants who received at least one dose of study drug. Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backward imputation were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 5-infected | Genotype 6-infected
Number analyzed (Participants) | 23 | 61
percentage of participants | 95.7 [79.0 to 99.2] | 98.4 [91.3 to 99.7]

2. Secondary Outcome: Percentage of Participants With On-treatment HCV Virologic Failure
Description: HCV virologic failure was defined as one of the following conditions:
  * confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < 15 IU/mL during the Treatment Period; or confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log10 IU/mL above nadir) at any time point during the Treatment Period; or
  * HCV RNA ≥ 15 IU/mL at end of treatment with at least 6 weeks of treatment, where the HCV RNA value must be collected on or after Study Drug Day 36 and study drug duration ≥ 36 days.
Time Frame: 8 or 12 weeks (depending on the treatment regimen)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 5-infected | Genotype 6-infected
Number analyzed (Participants) | 23 | 61
percentage of participants | 0.0 [0.0 to 14.3] | 1.6 [0.3 to 8.7]

3. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as confirmed HCV RNA ≥ 15 IU/mL between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment as planned with HCV RNA < 15 IU/mL at the end of treatment and had post-treatment HCV RNA data; participants who had been shown to be re-infected were not considered to have relapsed.
Time Frame: End of treatment (week 8 or 12 depending on the treatment regimen) through 12 weeks after the end of treatment.
Population: All enrolled participants who received at least one dose of study drug, with HCV RNA < 15 IU/mL at the end of treatment, at least one post-treatment HCV RNA value, and who completed the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 5-infected | Genotype 6-infected
Number analyzed (Participants) | 23 | 60
percentage of participants | 4.3 [0.8 to 21.0] | 0.0 [0.0 to 6.0]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug; 12 or 16 weeks depending on the treatment regimen.
Description: Adverse events are reported for the overall study population according to the prespecified analysis plan for this study.
Groups:
- Glecaprevir/Pibrentasvir: Participants received oral glecaprevir/pibrentasvir 300 mg/120 mg once daily for 8 or 12 weeks.
Arm/Group | Glecaprevir/Pibrentasvir
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 5/84
Other Adverse Events (participants affected / at risk) | 26/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=84)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ESCHERICHIA PYELONEPHRITIS (Infections and infestations) | 1 (1)
GASTRIC ULCER HELICOBACTER (Infections and infestations) | 1 (1)
GIARDIASIS (Infections and infestations) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=84)
NAUSEA (Gastrointestinal disorders) | 5 (5)
FATIGUE (General disorders) | 11 (11)
DIZZINESS (Nervous system disorders) | 6 (6)
HEADACHE (Nervous system disorders) | 11 (11)
INSOMNIA (Psychiatric disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT02966795/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02966795/SAP_001.pdf